CLINICAL TRIAL: NCT04390152
Title: Safety and Efficacy of Intravenous Infusion of Wharton's Jelly Derived Mesenchymal Stem Cell Plus Standard Therapy for the Treatment of Patients With Acute Respiratory Distress Syndrome Diagnosis Due to COVID 19: A Randomized Controlled Trial
Brief Title: Safety and Efficacy of Intravenous Wharton's Jelly Derived Mesenchymal Stem Cells in Acute Respiratory Distress Syndrome Due to COVID 19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Stopped by the IP, because the first 6 patients recruited had died and it was unknown if it represented any safety risk or if the sample was insufficient to evaluate the study hypotesis.
Sponsor: BioXcellerator (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIOXSOMCOV001
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: coronavirus; stem cell research; mesenchymal stem cell
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections | interventions — Hydroxychloroquine; Lopinavir; Ritonavir; Azithromycin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient code will be stored in sealed, opaque envelops with their respective codification. These envelops will be stored in Clinica Somer's Research Unit and the only person with access permission will be the pharmaceutical chemist in charge. Treatment delivery (MSC or placebo) will also be in charge of the chemist, guaranteeing blinding of patient and healthcare professionals. Data analysis will be done by people blind to the treatment received by each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell (Experimental): WJ MSC 50*10e6, two doses plus standard treatment with hydroxychloroquine + Lopinavir/Ritonavir or Azithromycin and ventilation support.
  Interventions: Drug: Wharton's jelly derived Mesenchymal stem cells.
- Control group (Active Comparator): Hydroxychloroquine, lopinavir/ritonavir and ventilation support plus placebo
  Interventions: Drug: Hydroxychloroquine, lopinavir/ritonavir or azithromycin and placebo (standard therapy)

INTERVENTIONS:
Drug: Wharton's jelly derived Mesenchymal stem cells. — IV Wharton's jelly derived Mesenchymal stem cells, two doses
  Arms: Mesenchymal stem cell
Drug: Hydroxychloroquine, lopinavir/ritonavir or azithromycin and placebo (standard therapy) — Standard therapy as per hospital protocol, hydroxychloroquine 400mg + Lopinavir/Ritonavir 400/100 or azithromycin 500mg and Placebo
  Arms: Control group

SUMMARY:
Recent COVID 19 pandemic has overwhelmed health services all around the world, and humanity has yet to find a cure or a vaccine for the treatment of patients, mainly the severe ones, who pose a therapeutic challenge to healthcare professionals given the paucity of information we have regarding SARS-CoV-2 pathogenesis.

Recently, reports mainly from China from patients treated with mesenchymal stem cells have shown promise in accelerating recovery, even in the critically ill and the therapy has sustained an increase in research because of it's powerful immunomodulatory effects, making it and interesting alternative in patients with lung and systemic inflammation.

These effects could help treat a lot of patients and improve their outcomes, reason why phase I/II studies are needed to show their safety and experimental efficacy.

DETAILED DESCRIPTION:
SARS-CoV-2, virus culprit of the COVID 19 that emerged in China, has become now a worldwide problem, with more than three million cases al around the world as reported by the World Health Organization. This situation has put health systems under extreme pressure, being overwhelmed be the amount of patients requiring attention.

Around 5% of patients will require ICU internation, due to severe lung inflammation giving rise to Acute Respiratory Distress Syndrome (ARDS) and a cytokine storm that ultimately affects other organs. In this group, mortality can be as high as 40%.

Mesenchymal stem cells (MSC) have shown great immunomodulatory effects, and are used in other inflammatory conditions as autoimmune diseases, being safe and preliminary effective in improving patients health status. They exert their effect via paracrine and autocrine pathways and have been shown to reduce IL-1, IL-6, Tumor necrosis factor alpha and increase IL-10 in COVID 19 patients. One of the greater advantages of the MSC is that they express no Major Histocompatibility Complex, reducing the risk of host immune reaction.

Given their immunomodulatory effects, research in this topic showing their safety and experimental efficacy are needed, as therapies for severe patients are lacking. Patients, researchers and data analysts will be blinded, and ARDS patients will be randomly allocated in standard therapy plus MSC arm or standard therapy alone to answer these questions.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 positive Real Time - Polymerase Chain Reaction
* Moderate to severe Acute respiratory distress syndrome according to Murray classification.
* PaO2/FiO2 less than 200 mmHg.
* Within 36 hours of orotracheal intubation.
* Absence of response with previous standard therapy.
* Willing to participate in the study expressed by patient or responsible caregiver.
* Not being in other clinical trial.

Exclusion Criteria:

* Current pregnancy.
* Cardiac rhythm abnormalities with instability.
* Acute congestive heart failure/cardiogenic shock.
* Severe comorbidities affecting mortality as defined by research group.
* Cancer history in the past 5 years.
* HIV, syphilis, hepatitis B or C.
* Concomitant use of immunosuppressive therapy with contraindication to MSC.
* Fivefold elevation of liver enzymes (ALT, AST).
* Chronic kidney disease with glomerular filtration rate below 30ml/min or dialytic needs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Intergroup mortality difference with treatment | 28 days.
  Evaluation of efficacy of WJ-MSC defined by mortality at 28 days of application.

SECONDARY OUTCOMES:
Number of patients with treatment related adverse events | 6 months.
  Safety evaluation of WJ-MSC describing and comparing incidence, type and severity of adverse events in both groups.
Difference in days of mechanical ventilation between groups | From ICU admission to 180 days.
  Evaluation of the effect of WJ-MSC in the time of mechanical ventilation compared between the two groups, as prolonged mechanical ventilation days are associated with higher complication risks as pneumonia, tracheostomy and death.
Median reduction of days of hospitalization | From hospital admission to 180 days.
  Evaluation of the effect of WJ-MSC in the time of hospitalization between the two groups as a measure of efficacy.
Median reduction of days of oxygen needs | From hospital admission to 180 days.
  Evaluation of the effect of WJ-MSC in the time of oxygen needs compared between the two groups as a measure of efficacy.
Difference between "Sequential Organ Failure Assessment" score between groups | Baseline to 7 days
  "Sequential Organ Failure Assessment" (SOFA) score is a tool used to determine the beginning and evolution of multiorgan failure, ranging from 0 to 24, being 24 the worst scenario. It has been proven useful as an outcome predictor of mortality and ICU stay. The result is the addition of the evaluation of each organ or system. Effect of WJ-MSC in the SOFA score will be compared between the two groups.
Difference between median Murray score between groups | Baseline and 7 days
  Murray score is a tool used to classify lung injury. 0 = no lung injury, 0.1-2.5, mild to moderate lund injury, >2.5 Acute respiratory distress syndrome.
  The effect of WJ-MSC in the Murray score will be compared between the two groups.
Difference in APACHE II score between groups | Baseline and 7 days
  APACHE II is a prognostic score based on 12 different items obtained in the first 24 hours of ICU admission. Its mainly used as a single measure, but some authors have used and described prediction usefulness with repeated measures. It ranges from 0 to 71 points. Higher scores are related to higher ICU mortality.
  The effect of WJ-MSC in the APACHE II score will compared between the two groups.
Difference in lymphocyte count between groups | baseline and 21 days or discharge
  Evaluation of the effect of WJ-MSC in lymphocyte count measured in absolute number/mm3.
  These laboratory measures have been associated with COVID 19 severity.
Changes in C reactive protein concentration between groups | baseline and 21 days or discharge
  Evaluation of the effect of WJ-MSC in C reactive protein concentration between the two groups, measured in mg/dl.
  Highest levels have been associated with COVID 19 severity and inflammation.
Changes in D dimer concentration | baseline and 21 days or discharge
  Evaluation of the effect of WJ-MSC in D dimer between the two groups, measured in micrograms Highest levels have been associated with COVID 19 severity and thromboembolic complications.
Changes in ferritin concentration | baseline and 21 days or discharge
  Evaluation of the effect of WJ-MSC in ferritin compared between the two groups, measured in nanograms/ml.
  These laboratory measures have been associated with COVID 19 infection and severity.
Changes in lactate dehydrogenase concentration | baseline and 21 days or discharge
  Evaluation of the effect of WJ-MSC in LDH compared between the two groups, measured in units/liter.
  These laboratory measures have been associated with COVID 19 infection and severity.
Impact on interleukin 6 concentrations between groups. | Baseline and 7 days
  Cytokines are biomarkers of inflammation or inflammatory activity in the human body. Changes in this profile give information about underlying process of inflammation.The effect of WJ-MSC in IL-6 will be compared between the two groups. It will be measured in picograms/ml.
Impact on interleukin 8 concentrations between groups. | Baseline and 7 days
  Cytokines are biomarkers of inflammation or inflammatory activity in the human body. Changes in this profile give information about underlying process of inflammation. The effect of WJ-MSC in IL 8 will be compared between the two groups. It will be measured in picograms/ml.
Impact on interleukin 10 concentrations between groups. | Baseline and 7 days
  Cytokines are biomarkers of inflammation or inflammatory activity in the human body. Changes in this profile give information about underlying process of inflammation. The effect of WJ-MSC in IL 10 will be compared between the two groups. It will be measured in picograms/ml.
Impact on tumor necrosis factor alpha concentrations between groups. | Baseline to 7 days.
  Cytokines are biomarkers of inflammation or inflammatory activity in the human body. Changes in this profile give information about underlying process of inflammation. The effect of WJ-MSC in TNF alpha will be compared between the two groups. It will be measured in nanograms/ml.

OTHER OUTCOMES:
Changes in 6 minute walk between groups | 6 months
  Evaluation of the effect of WJ-MSC in pulmonary function measured with 6 minute walk.
  6 minute walk is a test that gives information about pulmonary, cardiovascular and musculoskeletal functions. It measures the distance walked in 6 minutes in meters.
Changes in Pulmonary Computed Tomography Scan between groups | 6 months
  Evaluation of the effect of WJ-MSC in pulmonary function with thoracic CT scan. CT scan gives information about lung parenchyma, showing acute and chronic changes related to the underlying condition. Radiologic findings will be compared mainly comparing percentage of patients with pulmonary fibrosis.
Changes in Spirometry between groups | 6 months
  Evaluation of the effect of WJ-MSC in pulmonary function measured with spirometry, compared between the two groups. Spirometry gives information about lung volume and mobilization of air.
  Main parameters to be measured in spirometry are Forced Vital Capacity, Forced Expiratory Volume in 1 second and relation between these two to define if there is obstruction or restriction of airflow.
Changes in health related quality of life between groups | 6 months
  Evaluation of the effect of WJ-MSC in health related quality of life assessed by 36 Item Short Survey (SF-36).
  SF 36 is a patient reported tool. Each question is rated from 0 to 100, being 100 the best score possible. The scores are then compared to a population defined median score.
  Differences in global and specific scoring will be measured between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Hernandez-Ruiz, MSc, Principal Investigator — Clinica Somer
Locations (2):
- Colombia (2):
  - Clinical Somer, Rionegro, Antioquia
  - BioXcellerator, Medellín, Antioquia-CO

IPD SHARING:
Plan to Share IPD: No
Individual data won't be shared.